CLINICAL TRIAL: NCT06143358
Title: Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease With Qingkepingchuan Granules Clinical Observation of Phlegm-Heat and Lung Depletion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang Zhijie (Other)
Responsible Party: Sponsor-Investigator, Zhang Zhijie, PhD, Beijing University of Chinese Medicine
Organization: Beijing University of Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SY-1
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Qingkepingchuan Granules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Qingkepingchuan Granules+Conventional basic therapy
  Interventions: Drug: Qingkepingchuan Granules
- control subjects (Other): Conventional basic therapy
  Interventions: Other: conventional treatment

INTERVENTIONS:
Drug: Qingkepingchuan Granules — Qingkepingchuan Granules,Take it three times a day with water after meals.
  Arms: treatment group
Other: conventional treatment — Oxygen intake, selection of appropriate antibiotics based on lab results, and other treatments
  Arms: control subjects

SUMMARY:
Through the clinical observation of Qingcheng Pingxian Granules in the treatment of acute exacerbation of chronic obstructive pulmonary disease (phlegm-heat lung syndrome), (1) to evaluate the safety of Qingcheng Pingxian Granules in the acute exacerbation of chronic obstructive pulmonary disease; (2) to observe the clinical efficacy of Qingcheng Pingxian Granules in the treatment of acute exacerbation of chronic obstructive pulmonary disease, to provide an effective medication and solution for the treatment of acute exacerbation of chronic obstructive pulmonary disease, and to provide data for the development of the further application of Qingcheng Pingxian Granules.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of AECOPD.
2. Chinese medicine diagnosis is consistent with phlegm-heat and lung depletion evidence
3. 40 years old ≤ age ≤ 90 years old
4. Patients who signed the informed consent form and volunteered to participate in the study

Exclusion Criteria:

1. Combined with other primary lung diseases such as bronchial asthma, bronchiectasis, etc.
2. Combination of serious cardiovascular, urinary, digestive, haematopoietic, endocrine metabolic system diseases, other psychiatric and neurological diseases.
3. Pregnant or lactating patients.
4. Allergic to the clinical trial drugs.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Chinese Medicine Symptoms Scale | Before the start of treatment, 1 week of treatment, 2 weeks of treatment, 1 month of follow-up
  Record changes in patients' TCM indicators。The scale includes cough, wheezing, shortness of breath, sputum volume, chest tightness, sputum colour, sputum quality, fever, thirst, irritability, constipation, tongue coating, and pulse. The first four items are rated 0-6, and the last nine items are rated 0-3, with higher ratings indicating poorer treatment outcomes.
COPD assessment test | Before the start of treatment, 1 week of treatment, 2 weeks of treatment, 1 month of follow-up
  Record changes in the patient's condition
breathlessness measurement using the modified British Medical Research Council | Before the start of treatment, 1 week of treatment, 2 weeks of treatment, 1 month of follow-up
  Record changes in the patient's condition

SECONDARY OUTCOMES:
6-minute walking test | Before the start of treatment, 2 weeks of treatment
  Record changes in the patient's condition

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing University of Chinese Medicine, Beijing, China